CLINICAL TRIAL: NCT01773642
Title: Comparative Effectiveness of Pediatric HIV Disclosure Interventions in Uganda
Brief Title: Pediatric HIV Disclosure Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: MU-JHU CARE (Other)
Responsible Party: Principal Investigator, Lisa Butler, Associate Research Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pediatric HIV Disclosure
Record Dates: First submitted 2013-01-17; First posted 2013-01-23 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Paediatric HIV Diagnosis Disclosure
Keywords: pediatric HIV diagnosis disclosure; cognitive behavioral intervention; Uganda

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-behavioral intervention (Experimental): A cognitive-behavioural intervention aimed at supporting caregivers through paediatric HIV diagnosis disclosure to the child in their care.
  Interventions: Behavioral: Cognitive behavioral intervention to support pediatric HIV disclosure
- Standard of Care (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive behavioral intervention to support pediatric HIV disclosure
  Arms: Cognitive-behavioral intervention

SUMMARY:
With increased availability of antiretroviral therapy (ART) and improved care, increasing numbers of perinatally infected children are surviving into adolescence. While HIV care and treatment programs are expanding, growing challenge faced by health providers and caregivers is diagnosis disclosure to HIV infected children.

The investigators propose a 4 year project to test the effectiveness of a cognitive-behavioural intervention that the investigators have designed to support developmentally appropriate disclosure to HIV infected children by their caregiver.

The investigators hypothesize that the intervention will lead to increased disclosure rates and will over time improve health and mental health outcomes among caregivers and children in the intervention group compared to those receiving standard care. The findings of the study will inform Ugandan and other countries' national policies on pediatric HIV care and treatment.

DETAILED DESCRIPTION:
At the end of 2009, there were an estimated 2.1 million children < 15 years living with HIV, with almost 90% residing in sub-Saharan Africa (SSA). In Uganda alone there are an estimated 150,000 HIV-infected children. Although disclosing to a child that he or she is infected with HIV is an important and integral part of providing comprehensive HIV medical care, studies conducted in SSA have indicated that only 2% to 37.8% of HIV-infected children < 15 years know their HIV status. Studies by the investigators' team and others have revealed a high demand by both caregivers and children for health provider-facilitated communication about HIV and disclosure to HIV-infected children. In Uganda despite the rapid expansion of HIV services for children, very few health providers receive formal training in how to support disclosure of an HIV diagnosis to an infected child. Despite the existence of international and national recommendations for disclosure there are no tested models for supporting caregivers and HIV-infected children in SSA through the process of disclosure.

This study proposes to test the effectiveness of an innovative cognitive-behavioural intervention designed to support developmentally appropriate disclosure to HIV-infected children by their caregiver. The proposed intervention builds on the investigators' team's prior research is informed by a cognitive behavioral perspective, as well as the Disclosure Processes Model. The investigators will also adapt components of a multi-faceted program for caregivers of HIV-infected children, developed by members of the investigators' team with funding support from the US President's Emergency Plan for AIDS Relief (PEPFAR).

Specific aims:

1. To determine the effectiveness of a cognitive-behavior intervention for increasing disclosure of children's HIV diagnosis by caregivers to their HIV-infected children age 7-12 years old in Uganda.
2. To determine the effect of disclosure on immediate and longer-term caregiver and child mental health, and child behavioral and clinical outcomes, and whether the intervention modifies these effects
3. To assess the incremental cost, health impact, and cost-effectiveness of the intervention

ELIGIBILITY:
Inclusion criteria:

* children of age 7 to 12 years;
* confirmed HIV-infected;
* unaware of their HIV status, according to caregiver report;
* principal caregiver, age 18 years or older, of the eligible study child is able and willing to participate in their regular treatment program (monthly visits) and data collection visits at the study clinic at 6-month intervals for 24 months;
* agreement to participate in 3 group sessions with other caregivers over a 6 week period, and 3 counseling session with the eligible child(ren), scheduled at the same time as usual clinic visits;
* resides within a 30km radius around the study clinic, and not planning on moving during the study period; caregiver and child must both consent / assent for participation.

Exclusion criteria:

* caregivers and children who are unable to consent or assent to participation in the study due to cognitive impairment or illness;
* for children, medical history of serious birth complications, severe malnutrition, bacterial meningitis, encephalitis, cerebral malaria, or other known brain injury or disorder requiring hospitalization or continued evidence of seizure or other neurological disability;
* for caregivers, severe mental illness or developmental disability.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Disclosure to child of child's HIV-positive status | 24 months

SECONDARY OUTCOMES:
HIV related morbidity | 24 months
  For all children and HIV-infected caregivers, information on WHO stage of HIV infection, treatment status, opportunistic infections, CD4 counts will be abstracted from medical records.
Child antiretroviral medication adherence | 24 months
Cost and Cost-effectiveness | 24 months
Caregiver depression/anxiety | 24 months
Child behavior checklist | 24 months
  captures depression, anxiety and behavior using the child behavior checklist

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Butler, Principal Investigator — U Connecticut
Locations (6):
- Uganda (6):
  - Kampala City Council Authority (KCCA) Kiswa Health Centre, Kampala
  - KCCA Kawaala Health Centre, Kampala
  - KCCA Kisenyi Health Centre, Kampala
  - KCCA Kitebi Health Centre, Kampala
  - Makerere University-Johns Hopkins University Research Collaboration (MUJHU) clinic, Kampala
  - Nsambya Health Clinic, Kampala